CLINICAL TRIAL: NCT01592175
Title: Spatio-temporal Dynamic of the Relationship Between Spatial Attention and Visual Awareness
Brief Title: Magnetoencephalography (MEG), Attention and Conscience
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-49; 2011-A01554-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-04-16; First posted 2012-05-07 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Change in Sustained Attention; Awareness; Reaction Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The tight relationship between attention and conscious perception makes them difficult to study in isolation and has led many scientists to closely link these two processes. However, while some authors argue that conscious perception cannot occurs without attention, magnetoencephalography (MEG) and fMRI studies had shown that attention and consciousness are two distinct brain processes.

If endogenously triggered attention and consciousness are dissociated, it has been proposed that orienting of exogenous attention is a necessary, though not sufficient, antecedent of conscious perception.

In the present study we used MEG to explore the neural correlates of exogenous attention and consciousness during visual processing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 40 who have signed informed consent for participation to the study and are affiliated to a social security regimen
* right-handler, without auditory or visual deficit

Exclusion Criteria:

* history of neurological or psychiatic disease
* medication
* sensory disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults living in Paris or around fulfilling the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07-02 (Actual)

PRIMARY OUTCOMES:
Brain activity during visuo-spatial attention tasks | Three years
  Magnetoencephalography will be used to measured cerebral evoked potential and oscillatory activity, while subjects will performed a visuo-spatial attention task.

CONTACTS AND LOCATIONS:
Locations (1):
- CRICM, Paris, France